CLINICAL TRIAL: NCT06106399
Title: Ultrasound Guided Wide Awake Local Anesthesia Versus Clavipectoral Fascia Plane Block With Superficial Cervical Plexus Block for Clavicle Surgery, Prospective Randomized Clinical Trial
Brief Title: US Guided WALLANT vs CPB Block for Clavicle Surgery
Acronym: WALANT-CPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ismail Mohamed Abdelgawad Ahmed, DOCTOR, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WALANT-CPB in clavicle surgery
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Clavicle Fracture; Clavicle Injury
Keywords: wide awake local anesthesia; clavipectoral fascia plane block; clavicle surgery

STUDY DESIGN:
Intervention Model Description: 2 Arms model
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthiologist who perform postoperative pain will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WALLANT (group 1) (Active Comparator): wide awake local anesthesia and no tourniquet (WALLANT)
  Interventions: Procedure: WALLANT
- CPB (group 2) (Active Comparator): clavipectoral fascia plane block combined with superficial cervical plexus block (CPB)
  Interventions: Procedure: WALLANT

INTERVENTIONS:
Procedure: WALLANT — Comparison between (WALLANT) and (CPB) as a sole anesthesia in clavicle surgery
  Other Names: CPB

SUMMARY:
The clavicle is frequently fractured bone. regional anesthesia (RA) for clavicle surgery is always challenging due t complex innervation from the two plexuses (cervical and brachial). various RA techniques described for clavicle surgery include plexus blocks, fascial plane blocks,and truncal blocks.

DETAILED DESCRIPTION:
Clavipectoral Fascial Plane Block (CPB) is most commonly used as an anesthesia and postoperative analgesia technique to clavicle surgery.

This study is deigned to evaluate the feasibility of wide awake local anesthesia no tourniquet (WALANT) technique as a sole anesthesia in clavicle surgery, clavipectoral (CVP) fascia plane block + superficial cervical plexus plane block (CPB) as a sole anesthesia technique in clavicle surgery by using intraoperative verbal rating score (VRS) to determine how many patients need analgesia, sedation or convert to general anesthesia (GA), and postoperative assessment of patient satisfaction and 24 hour postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) 1,2
* Unilateral clavicle fracture.

Exclusion Criteria:

* psychologically unstable patient.
* uncooperative patient.
* patient refusal to be awake during surgery.
* allergy.
* infection at site of infection.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of the block as a sole anesthetic technique | 6 months
  intra-operative verbal rating score to determine how many patients need supplementary analgesia,sedation or converted to general anesthesia

SECONDARY OUTCOMES:
24 hour postoperative opioid consumption | 6 months
  Post-operative hourly VAS for the first 6 hours, at 8 hours, at 12 hours, at 16 hours,then at 24 hours postoperative
patient satisfaction | 6 months
  patient satisfaction score immediately postoperative on hospital discharge and after 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are planned to be coded for privacy protection

REFERENCES:
- [Background] Zhuo Q, Zheng Y, Hu Z, Xiong J, Wu Y, Zheng Y, Wang L. Ultrasound-Guided Clavipectoral Fascial Plane Block With Intermediate Cervical Plexus Block for Midshaft Clavicular Surgery: A Prospective Randomized Controlled Trial. Anesth Analg. 2022 Sep 1;135(3):633-640. doi: 10.1213/ANE.0000000000005911. Epub 2022 Jan 21. PMID 35061634
- [Background] Lee CCM, Beh ZY, Lua CB, Peng K, Fathil SM, Hou JD, Lin JA. Regional Anesthetic and Analgesic Techniques for Clavicle Fractures and Clavicle Surgeries: Part 1-A Scoping Review. Healthcare (Basel). 2022 Aug 7;10(8):1487. doi: 10.3390/healthcare10081487. PMID 36011144
- [Background] Azizi K, Benhamza S, Motiaa Y. Novel use of ultrasound guidance in wide-awake local anesthesia technique for clavicle surgery. Korean J Anesthesiol. 2022 Feb;75(1):103-105. doi: 10.4097/kja.21282. Epub 2021 Jun 30. No abstract available. PMID 35124948